CLINICAL TRIAL: NCT03462316
Title: To Evaluate the Efficacy of NY-ESO-1-specific T Cell Receptor (TCR) Affinity Enhancing Specific T Cell in Bone and Soft Tissue Sarcoma
Brief Title: NY-ESO-1-specific T Cell Receptor (TCR) T Cell in Sarcoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Xiangxue Precision Medical Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xing Zhang, Vice director of department of medical sarcoma and melanoma,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2017-023-01
Record Dates: First submitted 2018-01-16; First posted 2018-03-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Bone Sarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Bone Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NY-ESO-1 TCR Specific T cell Therapy (Experimental): NY-ESO-1 TCR specific T cells are prepared by lentiviral infection. Seven days before TCR-T cell reinfusion, the subjects received low-dose cyclophosphamide (15mg/kg/d x 3 days) and low-dose fludarabine (15mg/m2/d x 3 days) lymphocyte clearance. Four days later, TCR-T cells were transfused back (1 x 109-5 x 1010 was administered once or in stages). Then interleukin (IL)-2 subcutaneous injections (250,000 IU/twice/day) will be subcutaneously administered for 14 days concomitantly to each subject within 15-30 minutes after cell reinfusion. If the first three patients had no severe bone marrow suppression side effects (CTCAE was above grade 3) on low-dose lymphocyte clearance therapy, the dosage of cyclophosphamide (20 mg/kg/d x 3 days) and fludarabine (25 mg/m2/d x 3 days) could be increased for follow-up patients.
  Interventions: Biological: NY-ESO-1（TCR Affinity Enhancing Specific T cell Therapy）

INTERVENTIONS:
Biological: NY-ESO-1（TCR Affinity Enhancing Specific T cell Therapy） — NY-ESO-1（TCR Affinity Enhancing Specific T cell Therapy）

SUMMARY:
The main purpose of this trial is to investigate the safety and tolerability of NY-ESO-1（TCR Affinity Enhancing Specific T cell Therapy）in the first-line treatment failed advanced bone and soft tissue sarcoma. The secondary purpose of this trial is to investigate the efficacy of NY-ESO-1（TCR Affinity Enhancing Specific T cell Therapy）in the first-line treatment failed advanced bone and soft tissue sarcoma.

DETAILED DESCRIPTION:
This is a one arm, open label, dose escalation, single dose phase I study. The investigators include first-line treatment failed advanced patients with bone or soft tissue sarcoma and without standard regimen;TCR-T cell therapy has made a breakthrough for tumors in recent years. Phase I/II trial of NY-ESO-1-specific TCR-T treatment for synovial sarcoma and melanoma, conducted by the Rosenberg team at the National Cancer Institute, showed that 61% Synovial cell sarcoma patients and 55% melanoma patients benefit from this treatment, without severe side effects found in T cell receptor (TCR) transduced T-Cell Immunotherapy.

This clinical trial is mainly focused on cancer-testis antigen, because it is not expressed in normal cells. NY-ESO-1 antigen as one member of cancer-testis antigen, is commonly expressed in 10-50% of melanoma, lung, liver, esophageal, breast, prostate, bladder, thyroid and ovarian cancer cases, 60% of multiple myeloma cases, and 70-80% of synovial sarcoma. NY-ESO-1 expression was also found in 88.2% of myxoid liposarcomas, 61.1% of synovial sarcomas, 31.3% of osteosarcomas, 21.4% of pleomorphic liposarcomas, 16.7% of desmoplastic small round cell tumors, and 14.3% of chondrosarcomas. The NY-ESO-1 TCR cell therapy for synovial sarcoma and melanoma has benefited many patients, but its effect on bone and soft tissue sarcoma is still unknown. So the investigators plan to explore its efficacy.

The patients must meet the two criteria: HLA-A*0201+ and NY-ESO-1 positive cells≥25% by immunohistochemistry. By this trial, the dose-limiting toxicity (DLT) and maximum tolerance (MTD) will be initially identified.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent before undertaking any trial-related activities;
2. Aged 14 to 70 years old;
3. Patients withbone and soft tissue sarcoma in stage IV by licensed pathologist;
4. First-line treatment failed advanced patients.
5. With measurable lesions, the product of the two maximum vertical diameters should not be less than 5mm*5mm
6. Meet the two screening indicators: HLA-A*0201+, NYESO-1+(≥25% by immunohistochemistry);
7. Eastern Cooperative Oncology Group score 0-1; life expectancy is longer than 3 months;
8. The patient did not receive anti-tumor therapy within 4 weeks before enrollment;
9. A brain metastasis patient in a stable condition for one month after anti-tumor therapy can be included;
10. Left ventricular ejection fraction≥50%;
11. Lab test results meet the following requirements: white blood cell count≥3.0×10^9/L; absolute neutrophil count≥1.5 ×10^9/L (No human granulocyte colony stimulating factor support); absolute lymphocyte count≥0.7×10^9/L;blood platelet≥75 ×10^9/L; Hemoglobin≥10g/dL (No transfusion in the last 14 days); Prothrombin time or International normalized rate ≤1.5×normal upper limit, except taking anticoagulant therapy; thrombin time≤1.5×normal upper limit, except taking anticoagulant therapy; Serum creatinine: 1.5mg /dL (or 132.6 microns /L)；a 24-hour creatinine clearance rate≥60mL/ min; Aspartate transaminase / serum glutamic oxaloacetic transaminase≤2.5 ×upper limit of normal; Alanine aminotransferase/ serum glutamate pyruvate transaminase≤2.5 ×upper limit of normal; total bilirubin≤1.5×upper limit of normal.

    In the case of liver metastasis, glutamate transaminase and glutamate alanine transaminase should be less than 5 x ULN
12. Women of child-bearing age who have not undergone sterilization before menopause must agree to use effective contraceptive measures at least 30 days from the start of the study treatment to the last drug use, and serum pregnancy test is negative 14 days before the first treatment.
13. Men who have not received sterilization must agree to use effective contraception from the start of the study until at least 90 days after the last study medication is administered.
14. During the whole test period, the subjects can regularly go to the enrolled research institutions for relevant detection, evaluation and management.

Exclusion Criteria:

1. other types of tumors; If the patient has a previous history of malignant tumor, the disease-free time of the patient needs > for 5 years.
2. received major surgery, conventional chemotherapy, large-area radiotherapy, immune therapy or any biological anti-tumor therapy within 4 weeks before enrollment;
3. allergic to ingredients in this trial;
4. common terminology criteria for adverse events not return to under 2 level from previous surgery or treatment-related adverse reactions;
5. poorly managed hypertension (systolic blood pressure >160 mmHg and / or diastolic blood pressure > 90 mmHg) or clinically serious (for example, active) cerebrovascular diseases such as cerebrovascular incident (within 6 months prior to signing the informed consent), myocardial infarction (within 6 months prior to signing the informed consent), unstable angina, grade II or above heart failure according to New York Heart Association Grading Congestive, or severe arrhythmia can not be controlled by medication or has a potential impact on the study; with consecutive three times of obvious abnormality on electrocardiogram or average QT corrected interval ≥450 millisecond;
6. combined with other serious organic and mental disorders;
7. serious or active bacteria, viral or fungal infections that require systemic treatment;
8. with autoimmune diseases: such as a history of inflammatory bowel disease or other autoimmune diseases determined by the investigator as unsuitable for the study (e.g. systemic lupus erythematosus,vasculitis, invasive pulmonary disease);
9. within 4 weeks prior the infusion, received chronic systemic steroid cortisone, hydroxyurea, immunomodulatory treatment (for example: Interleukin 2, alpha or gamma interferon, granulocyte colony stimulating factor, mammalian target of rapamycin inhibitors, cyclosporine, Thymosin etc);
10. with organ transplantation, autologous/allogeneic stem cell transplantation and renal replacement therapy;
11. with uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or liver failure;
12. alcohol and / or drug abuse;
13. pregnant or lactating women;
14. with any medical condition or disease determined by the investigators that may be detrimental to this trial;
15. without legal capacity / limited behavior.
16. receive any other gene therapy products before study

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v3.0 | 270 days
  safety evaluation(dose-limiting toxicity and the maximum tolerance)

SECONDARY OUTCOMES:
clinical response rate | 270 Days
  Overall Response Rate as assessed by RECIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Univerisity, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903